CLINICAL TRIAL: NCT07110857
Title: Evaluation of the Superficial Cervical Plexus Block in Oncological Throat and Neck Surgery
Acronym: BCS-ORL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP230866; PHRCI-2022-38 (Other Grant/Funding Number: Ministry of health, France); 2024-510942-15-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-25; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: ENT Cancers
Keywords: the superficial cervical plexus block; surgery; locoregional anesthesia; locoregional analgesia; ENT surgery
MeSH Terms: interventions — Cervical Plexus Block; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naropeine Arm (Experimental): Superficial cervical plexus block with 0.2 % ropivacaine (Naropeine)
  Interventions: Procedure: Cervical plexus block with 0.2 % Naropeine
- Placebo Arm (Placebo Comparator): Superficial cervical plexus block with 0.9 % saline placebo
  Interventions: Procedure: Cervical plexus block with saline placebo

INTERVENTIONS:
Procedure: Cervical plexus block with 0.2 % Naropeine — Under ultrasound guidance, a superficial cervical plexus block is performed immediately after induction and before skin incision by injecting 15-25 mL of 0.2 % ropivacaine (Naropeine) uni- or bilateral depending on the surgical incision
  Arms: Naropeine Arm
Procedure: Cervical plexus block with saline placebo — Under ultrasound guidance, a superficial cervical plexus block is performed immediately after induction and before skin incision by injecting 15-25 mL of 0.9 % saline uni- or bilateral depending on the surgical incision
  Arms: Placebo Arm

SUMMARY:
This national, prospective, multicenter, randomized study aims to reduce the amount of intravenous morphine (titration + PCA morphine) during the first 24 postoperative hours via a locoregional anesthesia technique in patients undergoing throat and neck cancer surgery.

DETAILED DESCRIPTION:
The incidence of throat and neck (ENT) cancers is 15000 new cases/year in France. Nowadays, there are no studies with a sufficient level of evidence to establish formal recommendations on analgesic treatments to be applied in the context of ENT cancer surgery.

As cancer surgery causes severe acute postoperative pain and chronic pain, loco-regional anesthesia (LRA) plays an increasingly role in the prevention of this type of pain.

However, nowadays there is no data in the literature highlighting the interest of LRA in the context of ENT cancer surgery, despite a significant theoretical benefit.

The superficial cervical block, already used in carotid or thyroid surgery, has already shown its value. It seems logical to propose this block in throat and neck cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient undergoing ENT cancer surgery with cervicotomy
* Adult patient having received oral information from a doctor and signed written consent
* Affiliation to a social security scheme, Universal Medical Coverage (CMU)

Exclusion Criteria:

* Patient refusal
* Altered mental faculties or patient unable to give consent
* Allergy to local anesthetics
* Severe respiratory pathology (altered respiratory function tests with 50% < FEV1 < 80%, FEV1/FVC < 70%, COPD stage 2 or more)
* Preoperative SpO2 less than 92% in ambient air
* Left heart failure NYHA 3 or more, impaired LVEF < 30% or less
* Lower respiratory infection in the month preceding surgery
* History of ENT cancer surgery with cervical lymph node dissection
* Pregnant or breastfeeding woman
* Patient under AME
* Patient under guardianship or reinforced curatorship
* Participation in other interventional research

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Amount of morphine | The first 24 hours postoperatively
  The analysis metric is the cumulative amount of IV morphine (amount of morphine titrated in SSPI + administered by PCA in mg and mg/kg/day) during the first 24 hours postoperatively.

SECONDARY OUTCOMES:
Remifentanil consumption | Intraoperative
  Change in remifentanil consumption during surgery per unit time (in µg/kg/min). The analysis metric is the cumulative sum of intraoperative remifentanil during surgery.
Consumption of morphine | In the first 72 hours postoperatively
  Change in consumption of morphine equivalent intravenous or oral in the first 72 hours postoperatively (mg and mg/kg). The analysis metric is the cumulative amount of morphine administered during the first 72 hours postoperatively.
Evaluation in cervical VAS and flap site VAS score | On arrival, 1 hour later, 2 hours later, 4 hours later
  Change in cervical VAS (Visual Analog Scale) and flap site VAS score in PACU (post anesthesia care units). The VAS measures pain intensity on a scale from 0 to 10, with two end points representing 0 'no pain' and 10 'pain as bad as it could possibly be'. The analysis metric is the change from baseline.
Evaluation in cervical VAS in dynamic conditions and flap site VAS score | Day 1, day 15 (or hospital discharge), 1 month and 3 months
  Change in cervical VAS (Visual Analog Scale) in dynamic conditions and flap site VAS score. The VAS measures pain intensity on a scale from 0 to 10, with two end points representing 0 'no pain' and 10 'pain as bad as it could possibly be'. The analysis metric is the change from baseline.
DN4 score assessment | Day 1, Day 15 (or hospital discharge), 1 month and 3 month
  DN4 (Douleur Neuropathique 4) score change. When the practitioner suspects neuropathic pain, the DN4 questionnaire is a useful diagnostic tool. If the patient's score is equal to or greater than 4/10, the test is positive indicating the presence of neuropathic pain. The analysis metric is the final value.
Evaluation of adverse effects attributable to morphine consumption | Day 1, Day 15 (or hospital discharge)
  Report / Change of adverse effects attributable to morphine consumption (desaturation, nausea-vomiting, etc.). The analysis metric is the difference between the post-processing value and the initial value.
Evaluation of the rate of patients with early rehabilitation | Initiated on Day 1
  Change in the rate of patients with early rehabilitation: standing, wheelchair, physiotherapy
The length of time spent in hospital | Duration of hospital stay assessed up to 15 days or hospital discharge
  Reduction in the length of hospitalization between the control arm and the experimental arm. The analysis metric is the final value.
Evaluation of the E Satis MSO FNAH score | Day 15 (or hospital discharge)
  Improvement of the E-Satis MSO (medical-surgery-obstetrics) FNAH (French National Authority for Health) score. E-Satis is expressed out of 100. Score close to 100: positive experience
Evaluation of the Mc Gill Pain score (SF-MPQ-2) | Day 1, day 15 (or hospital discharge), 1 month and 3 months
  Improvement in Mc Gill Pain score (SF-MPQ-2). The McGill Pain Index is a self-assessment scale that describes the quality and intensity of pain from 0 to 50. A score close to 50 indicates extremely severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia Desplanque, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (7):
- France (7):
  - CHU de Lille- Hôpital Roger Salengro, Lille
  - Assistance publique - Hôpitaux de Marseille, Marseille
  - AP-HP - Hôpital Lariboisière, Paris
  - Assistance publique - Hôpitaux de Paris, Paris
  - CHU Charles Nicolle, Rouen
  - hôpital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with European General Data Protection Regulation (GDPR).